CLINICAL TRIAL: NCT07240116
Title: An Open-Label, Randomized, 3-Treatment, 3-Period, 6-Sequence, Balanced Crossover Study to Characterize the Relative Bioavailability of Miricorilant Administered as 50-mg and 100-mg Kinetisol Tablets vs the 50-mg Spray Dried Dispersion Tablet Formulation With an Optional Food Effect Assessment in Healthy Adult Subjects
Brief Title: Study Evaluating the Bioavailability of Miricorilant With Optional Food Effect Assessment in Healthy Adult Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CORT118335-859
Record Dates: First submitted 2025-11-07; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — CORT118335

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Miricorilant Treatment Sequence A, B, C (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment A; in Period 2, treatment B; in Period 3, treatment C. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Miricorilant Treatment Sequence B, C, A (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment B, in Period 2, treatment C; in Period 3, treatment A. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Miricorilant Treatment Sequence C, A, B (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment C; in Period 2, treatment A; in Period 3, treatment B. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Miricorilant Treatment Sequence B, A, C (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment B; in Period 2, treatment A; in Period 3, treatment C. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Miricorilant Treatment Sequence A, C, B (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment A; in Period 2, treatment C; in Period 3, treatment B. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Miricorilant Treatment Sequence C, B, A (Experimental): Participants will receive a single dose of study drug in a fed state on Day 1 of each of 3 treatment periods. In Period 1, treatment C; in Period 2, treatment B; in Period 3, treatment A. A washout period of at least 7 days will follow each dose of the study drug.
  Interventions: Drug: Miricorilant Treatment A; Drug: Miricorilant Treatment B; Drug: Miricorilant Treatment C
- Optional Miricorilant Treatment D (Experimental): After completion of Period 3, analysis of pharmacokinetic and safety data will be used to decide if Period 4 will be conducted. In Period 4, selected participants will receive a single dose of treatment D in a fasted state on Day 1.
  Interventions: Drug: Miricorilant Treatment D

INTERVENTIONS:
Drug: Miricorilant Treatment A — Miricorilant 100 mg (1 x 100 mg) Kinetisol immediate release (IR) tablet for oral administration
  Other Names: CORT118335
  Arms: Miricorilant Treatment Sequence A, B, C; Miricorilant Treatment Sequence A, C, B; Miricorilant Treatment Sequence B, A, C; Miricorilant Treatment Sequence B, C, A; Miricorilant Treatment Sequence C, A, B; Miricorilant Treatment Sequence C, B, A
Drug: Miricorilant Treatment B — Miricorilant 100 mg (2 x 50 mg) Kinetisol IR tablet for oral administration
  Other Names: CORT118335
  Arms: Miricorilant Treatment Sequence A, B, C; Miricorilant Treatment Sequence A, C, B; Miricorilant Treatment Sequence B, A, C; Miricorilant Treatment Sequence B, C, A; Miricorilant Treatment Sequence C, A, B; Miricorilant Treatment Sequence C, B, A
Drug: Miricorilant Treatment C — Miricorilant 100 mg (2 x 50 mg) SDD IR tablet for oral administration
  Other Names: CORT118335
  Arms: Miricorilant Treatment Sequence A, B, C; Miricorilant Treatment Sequence A, C, B; Miricorilant Treatment Sequence B, A, C; Miricorilant Treatment Sequence B, C, A; Miricorilant Treatment Sequence C, A, B; Miricorilant Treatment Sequence C, B, A
Drug: Miricorilant Treatment D — Miricorilant 100 mg (1 x 100 mg or 2 x 50 mg) Kinetisol IR tablet for oral administration. The tablet strength administered will be decided after Period 3 is complete.
  Other Names: CORT118335
  Arms: Optional Miricorilant Treatment D

SUMMARY:
This single-center, randomized, open-label study will assess the relative bioavailability of 2 miricorilant (CORT118335) tablet formulations.

DETAILED DESCRIPTION:
This study will evaluate relative bioavailability of Kinetisol and spray dried dispersion (SDD) miricorilant (CORT118335) tablets. This study will consist of 6 possible treatment sequences across 3 periods for healthy, fed participants. A fourth period may be added to assess the impact of fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand written informed consent
* Willing and able to comply with study requirements
* Willing to comply with protocol-specified contraception requirements
* Healthy male or non-pregnant, non-lactating female of non-childbearing potential per Investigator assessment.
* Body mass index (BMI) of 18.0 to 30.0 kg/m^2 at screening
* Weight of at least 50 kg at screening

Exclusion Criteria:

* Serious adverse reaction or hypersensitivity to any drug or formulation excipients
* History of clinically significant allergy requiring treatment
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal (GI) disease, neurological or psychiatric disorder
* Any form of cancer within the 5 years before the first does of this study
* History and/or symptoms of adrenal insufficiency
* History of clinically significant GI disease
* Condition or history of a condition that could be aggravated by glucocorticoid antagonism or glucocorticoid activation
* History of additional risk factors for torsades de pointes
* Poor venous access that limits phlebotomy
* Clinically significant abnormal clinical chemistry, hematology or urinalysis
* History or evidence of hypokalemia
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
* Evidence of renal impairment at screening
* Positive serum or highly sensitive urine pregnancy test at screening or first admission
* Clinically significant ECG abnormalities or vital sign abnormalities at screening or baseline
* Received any investigational medicinal products (IMP) in a clinical research study within 5 half-lives or within 30 days prior to first dose
* Donation of blood within 2 months or donation of plasma within 1 week prior to first dose of study medication
* Are taking, or have taken, any prescribed or over-the-counter drug or vitamins/herbal remedies in the 14 days before first IMP administration
* Currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months before first IMP administration or 3 months for inhaled products
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption as defined in the study protocol
* A confirmed positive alcohol urine test at screening or first admission
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* A confirmed positive urine cotinine test at screening or first admission
* Positive drug screen test result at screening or first admission
* Male subjects with pregnant or lactating partners
* Study site or Sponsor employee or immediate family members one
* Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Time of Maximum Observed Concentration (Tmax) of Miricorilant | Predose and at serial timepoints up to 72 hours postdose
Maximum Observed Concentration (Cmax) of Miricorilant | Predose and at serial timepoints up to 72 hours postdose
Concentration at 24 Hours Postdose (C24) of Miricorilant | Predose and at serial timepoints up to 24 hours postdose
Area Under the Curve from Time 0 to the Time of Last Measurable Concentration (AUC[0-last]) of Miricorilant | Predose and at serial timepoints up to 72 hours postdose
Area Under the Curve from Time 0 Extrapolated to Infinity (AUC[0-inf]) of Miricorilant | Predose and at serial timepoints up to 72 hours postdose
Terminal Elimination Half-Life (T1/2) of Miricorilant | Predose and at serial timepoints up to 72 hours postdose
Relative Bioavailability (Frel) for Miricorilant Based on Cmax | Predose and at serial timepoints up to 72 hours postdose
Frel for Miricorilant based on AUC(0-last) | Predose and at serial timepoints up to 72 hours postdose
Frel for Miricorilant Based on AUC(0-inf) | Predose and at serial timepoints up to 72 hours postdose

SECONDARY OUTCOMES:
Number of Participants with Abnormal, Clinically Significant Clinical Laboratory Findings | Day -1 and 72 hours postdose in periods 3 and 4
  Clinical laboratory findings include hematology, clinical chemistry, urinalysis.
Number of Participants with Abnormal, Clinically Significant 12-Lead Electrocardiogram (ECG) Findings | Day -1, predose, and at 4 and 72 hours postdose in every study period
Number of Participants with Abnormal, Clinically Significant Vital Sign Findings | Day -1, predose, and at serial time points up to 72 hours postdose in every study period
Number of Participants with Abnormal, Clinically Significant Physical Exam Findings | 72 hours postdose in periods 3 and 4
Number of Participants with 1 or More Adverse Events | Screening up to 30 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No